CLINICAL TRIAL: NCT07217847
Title: Testing a Single-session Consultation for Reducing Binge Eating
Brief Title: Testing SHAPE: A Single-Session Intervention Targeting Binge Eating in Women Through Assessment and Values-Based Strategies
Acronym: SHAPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taylor Rezeppa (Other)
Collaborators: Ohio University (Other)
Responsible Party: Sponsor-Investigator, Taylor Rezeppa, Doctoral Candidate in Clinical Psychology, Ohio University
Organization: Ohio University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-FY26-100
Record Dates: First submitted 2025-10-14; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Binge Eating; Binge Eating Behaviour; Binge Eating/Loss of Control Eating; Body Image; Body Image Disturbance
Keywords: single session; single-session consultation; single-session intervention; binge eating; disordered eating; binge-spectrum disorder; body image; body image concerns; weight/shape concerns; overvaluation; loss of control eating
MeSH Terms: conditions — Bulimia; Binge-Eating Disorder; Body Weight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Assessment-only (Active Comparator): Diagnostic items of the Eating Disorder Examindation (EDE)
  Interventions: Behavioral: Assessment-only
- Full Intervention (SHAPE) (Active Comparator): Diagnostic items of the Eating Disorder Examindation (EDE)
  + Values-based reflection and goal-setting exercises
  Interventions: Behavioral: Assessment-only; Behavioral: values-based reflection and goal-setting/action-planning exercises
- Minimal-Assessment Control (Placebo Comparator): Intro/Eating Pattern + Bulimic Episodes/Overeating Sections of Eating Disorder Examindation (EDE)
  Interventions: Behavioral: Minimal-Assessment Control

INTERVENTIONS:
Behavioral: Assessment-only — Diagnostic items of the Eating Disorder Examindation (EDE)
  Arms: Assessment-only; Full Intervention (SHAPE)
Behavioral: values-based reflection and goal-setting/action-planning exercises — Assessment-only intervention + values-based reflection and goal-setting/action-planning exercises
  Other Names: SHAPE
  Arms: Full Intervention (SHAPE)
Behavioral: Minimal-Assessment Control — Invovles completing only the Intro/Eating Pattern + Bulimic Episodes/Overeating Sections of Eating Disorder Examination (EDE)
  Arms: Minimal-Assessment Control

SUMMARY:
The goal of this controlled trial is to learn whether a brief single-session intervention (SSI) can reduce binge eating symptoms by targeting overvaluation of weight/shape in women with recurrent binge eating.

The main questions it aims to answer are:

* Does assessment alone reduce binge eating severity and overvaluation of weight/shape compared to a control group undergoing minimal assessment?
* Does adding a values-based reflection and goal-setting component (the full SHAPE intervention) add benefits beyond the assessment alone?

Researchers will compare three groups:

1. assessment-only,
2. full SHAPE intervention, and
3. minimal assessment control to see if both active conditions outperform the control, and whether the full intervention adds any benefits beyond the assessment itself

Participants will:

* Complete a semi-structured eating disorder assessment (Eating Disorder Examination)
* Depending on assignment, also complete a values-based reflection and goal-setting exercise with psychoeducation
* Complete follow-up assessments evaluating binge eating severity, overvaluation of weight/shape, clinical impairment, binge frequency, and related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Identify as cisgender female
* self-reported BMI ≥ 18.5 kg/m²
* Rate the extent to which their weight or shape influences how they feel about themselves as a "4" or higher on a 7-point Likert scale on screening measures
* ≥1 binge eating episode every 2 weeks (i.e., ≥ six episodes over 3 months) at the time of screening

Exclusion Criteria:

* < 18 years old
* Assigned male at birth
* Gender identity different from biological sex indicated on birth certificate
* Purging behaviors (i.e., self-induced vomiting, laxative misuse, or diuretic misuse) ≥ 1x/week in the last 3 months at the time of screening.
* Engaged in structured psychological therapy or counseling (defined as attending sessions > 1x/month in the past 3 months)
* Prior participation in studies that include administration of the EDE interview at Ohio University (IRB-FY24-403, IRB-FY25-330, and IRB-21-F-14).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender female
Enrollment: 56 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Changes in overvaluation of weight/shape | 1 month
  Changes in Shape/weight overvaluation subscale score on 7-Item Eating Disorder Examination Questionnaire
Change in binge eating severity | 1 month
  Change in scores on Binge Eating Scale

SECONDARY OUTCOMES:
Change in Body Image Flexibility | 1 month
  5-item Body Image Acceptance and Action Questionnaire
Change in eating self-efficacy | 1 month
  Score change on Eating Self-Efficacy Brief Scale
Change in readiness to change eating disorder symptoms | 1 month
  Change in Eating Disorder Readiness Ruler scores
Change in eating disorder-related clinical impairment | 1 month
  Score change on Clinical Impairment Assessment
Change in depressive symtpoms | 1 month
  Change in Patient Health Questionnaire-8 scores
Change in binge eating frequency | 1 month
  Change in binge episode count on Eating Disorder Examination Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Katherine J. Forney, Ph.D., Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided